CLINICAL TRIAL: NCT06633913
Title: Neural Effects of Transcranial Magnetic Stimulation Using Concurrent Functional Magnetic Resonance Imaging
Brief Title: Concurrent TMS-fMRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jing Jiang (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Jing Jiang, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202402416; R01MH136197 (NIH)
Record Dates: First submitted 2024-09-30; First posted 2024-10-09 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Healthy Control; Depression; Anxiety
Keywords: Depression; Anxiety; TMS; fMRI; TMS-fMRI; TBS; Functional Connectivity; Individual Differences; Mood Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- spTMS-TBS-spTMS (Experimental): This is an open-label, single-arm study. The intervention will be delivered in spTMS-TBS-spTMS order to the dorsolateral prefrontal cortex (dlPFC) and vertex for each participant as described in the "Interventions" section. The order of the stimulation sites will be counterbalanced across participants.
  Interventions: Device: spTMS-TBS-spTMS

INTERVENTIONS:
Device: spTMS-TBS-spTMS — This study uses fMRI in combination with single-pulse TMS (spTMS) and theta-burst stimulation (TBS) to determine if the two effects coming from each are related to one another, and if there will be changes in brain activity when undergoing spTMS that are induced by TBS. Additionally, by stimulating the dlPFC in both patients and healthy controls with this paradigm, researchers are able to specifically compare the after-TBS single-pulse TMS-evoked brain responses with before-TBS responses to observe if TBS will change neural pathways disrupted in those who display high negative affect (e.g. depression, anxiety).

SUMMARY:
The goal of this clinical trial is to examine the neural mechanisms underlying transcranial magnetic stimulation (TMS) using concurrent functional magnetic resonance imaging (fMRI) in both healthy controls (HCs) and patients with high negative affect symptoms, such as depression and anxiety. Approximately half male and half female participants aged 18-65 will be recruited.

The main questions it aims to answer are:

1. Is the acute/transient effect induced by single-pulse TMS related to the long-term modulatory effect induced by repetitive TMS (rTMS)?
2. Do any of these effects predict negative affect symptoms, such as depression and anxiety?

Participants will:

1. Complete several tests to assess their cognitive abilities and emotional states
2. Undergo several brain scans, including resting-state fMRI, structural MRI, diffusion tensor imaging (DTI), and task fMRI
3. Have two different types of TMS sequences, single-pulse and repetitive pulses, administered to specific brain regions while undergoing fMRI

DETAILED DESCRIPTION:
The purpose of this study is to examine the neural mechanisms underlying transcranial magnetic stimulation (TMS) using concurrent functional magnetic resonance imaging (fMRI). Research is conducted in both healthy controls (HCs) and patients with high negative affect symptoms, such as depression and anxiety. Participants will undergo two visits, the first lasting about two hours and the second, scheduled within one week of the first, lasting about one hour. Approximately half male and half female participants aged 18-65 will be recruited. The aims are to examine (1) whether the acute/transient effect induced by single-pulse TMS is related to the long-term modulatory effect induced by rTMS, and (2) whether any of these effects predict negative affect symptoms, such as depression and anxiety.

In the first visit, participants will complete several tests to assess their cognitive abilities and emotional states, specifically measuring depression and anxiety levels. These tests will help explore the relationship between their cognitive/emotional states and brain activity during TMS-fMRI. After the tests, participants will undergo several brain scans to determine the best locations for TMS during the second visit and to measure the strength of connections between different brain regions. During the second visit, participants will undergo three parts of TMS-fMRI scanning. The first part involves applying single-pulse TMS to the dorsolateral prefrontal cortex (DLPFC) and a control area (the vertex) while taking fMRI scans. This helps elucidate how TMS affects deep brain regions related to mood disorders. By comparing brain responses to TMS between healthy controls and patients, researchers can gain important knowledge of whether the neural pathways between stimulated region and these subcortical brain regions are disrupted in patients. The second part includes theta-burst stimulation (TBS) of TMS to the DLPFC, which is a stimulation protocol approved by Food and Drug Administration (FDA). Finally, in the third part, single-pulse TMS is administered again after TBS to see if the TBS has changed the brain's response. Comparing the after-TBS single-pulse TMS-evoked brain responses with before-TBS responses would allow the investigators to track whether the TBS could change the disrupted neural pathways in patients. Investigators will also examine how participants' cognitive/emotional test results and brain connectivity relate to the TMS-evoked brain responses and the effects of TBS. Any potential relationships found can provide insight into the underlying mechanisms of how individual differences in cognitive/emotional functioning and brain connectivity profile might influence or be influenced by brain stimulation, which could ultimately inform personalized approaches to neuromodulation therapies.

ELIGIBILITY:
Inclusion for patients:

* Diagnosis of major depressive disorder and/or general anxiety disorder
* Age greater than or equal to 18 years
* Age less than or equal to 65 years
* Able to understand and consent for research participation
* English-speaking

Inclusion for healthy controls:

* Report no lifetime psychiatric diagnosis and treatment
* scores on Patient Health Questionnaire (PHQ-9) and Generalized Anxiety Disorder Questionnaire (GAD-7) lower than 4
* Age greater than or equal to 18 years
* Age less than or equal to 65 years
* Able to understand and consent for research participation
* English-speaking

Exclusion for all subjects:

* Age less than 18 years
* Age greater than 65 years
* With epilepsy or seizure disorder
* With implanted ferromagnetic equipment in their face or skull near the stimulation target

MRI Exclusion criteria for all subjects:

* Implanted device including pacemaker, coronary stent, defibrillator, or neurostimulation device that is not MRI-compatible
* Metal in body including bullets, shrapnel, metal slivers
* Claustrophobia
* Uncontrolled high blood pressure
* Blood circulation problems
* Opiate medication, antihypertensive medication, or any medication that interferes with blood flow (interferes with fMRI recordings)
* Significant heart disease, such as atrial fibrillation
* Pregnancy in female participants
* Prior exposure to deep brain stimulation, rTMS, or tDCS (transcranial direct current stimulation) therapies
* History of neurological or cardiovascular disorders, brain surgery, radiation treatment, brain hemorrhage or tumor, stroke, or diabetes
* Significant traumatic brain injury (loss of consciousness, post-injury amnesia, significant radiological/neurological findings, penetrating brain injury)
* Refusal to abstain from illicit drug use for duration of the study
* Refusal to abstain from alcohol within 24 hours of scans

If you would like to participate in the study, click this link to fill out the Screening Form: https://redcap.icts.uiowa.edu/redcap/surveys/?s=DEYHWF8TMCHHW4Y7

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Pre and Post TBS Modulation Effect Comparison | Up To 10 Minutes
  The primary outcome measure will be the modulation effect of TBS to the dlPFC, which is the difference between TMS-induced acute/transient effects before and after TBS. The acute/transient effects will be assessed through single-pulse TMS-induced fMRI blood oxygenation level-dependent (BOLD) responses. The difference in BOLD response before and after TBS (i.e., TBS modulation effect) will be assessed using paired t-tests reported with t and p values.
Difference in TBS Modulation Effect Across Comparison Groups | Up to 10 Minutes
  Another primary outcome measure is whether this TBS modulation effect is different between healthy controls and patients with high negative affect symptoms (e.g. depression, anxiety). The difference will be assessed using independent t-tests reported with t and p values.

SECONDARY OUTCOMES:
TMS Effects with Neurocognitive and Emotion Functions | One Week
  The secondary outcome measure is the relationship between the TBS modulation effect, TMS-induced acute/transient effects, intrinsic network properties, and participants' neurocognitive and emotion functions. This relationship will be assessed using the Pearson correlation reported using r and p values.
  The intrinsic network properties will be assessed by participants' (1) resting-state fMRI-based functional connectivity reported with Pearson based r values between two brain regions, (2) DTI MRI-based structural connectivity reported by the number of white matter streamlines. The neurocognitive functions will be assessed with cognitive scales and questionnaires (e.g. Montreal Cognitive Assessment (MOCA)). The emotion functions will be assessed emotional scales and questionnaires (e.g. Montgomery-Åsberg Depression Rating Scale (MADRS)).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Carver College of Medicine, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be submitted to the NIMH Data Archive every 6 months.

REFERENCES:
- [Background] Mueller JK, Grigsby EM, Prevosto V, Petraglia FW 3rd, Rao H, Deng ZD, Peterchev AV, Sommer MA, Egner T, Platt ML, Grill WM. Simultaneous transcranial magnetic stimulation and single-neuron recording in alert non-human primates. Nat Neurosci. 2014 Aug;17(8):1130-6. doi: 10.1038/nn.3751. Epub 2014 Jun 29. PMID 24974797
- [Background] Kobayashi M, Pascual-Leone A. Transcranial magnetic stimulation in neurology. Lancet Neurol. 2003 Mar;2(3):145-56. doi: 10.1016/s1474-4422(03)00321-1. PMID 12849236
- [Background] Khedr EM, Rothwell JC, Ahmed MA, El-Atar A. Effect of daily repetitive transcranial magnetic stimulation for treatment of tinnitus: comparison of different stimulus frequencies. J Neurol Neurosurg Psychiatry. 2008 Feb;79(2):212-5. doi: 10.1136/jnnp.2007.127712. PMID 18202212
- [Background] Hosomi K, Shimokawa T, Ikoma K, Nakamura Y, Sugiyama K, Ugawa Y, Uozumi T, Yamamoto T, Saitoh Y. Daily repetitive transcranial magnetic stimulation of primary motor cortex for neuropathic pain: a randomized, multicenter, double-blind, crossover, sham-controlled trial. Pain. 2013 Jul;154(7):1065-72. doi: 10.1016/j.pain.2013.03.016. Epub 2013 Mar 15. PMID 23623156
- [Background] George MS. Whither TMS: A One-Trick Pony or the Beginning of a Neuroscientific Revolution? Am J Psychiatry. 2019 Nov 1;176(11):904-910. doi: 10.1176/appi.ajp.2019.19090957. PMID 31672044
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Blumberger DM, Fitzgerald PB, Mulsant BH, Daskalakis ZJ. Repetitive transcranial magnetic stimulation for refractory symptoms in schizophrenia. Curr Opin Psychiatry. 2010 Mar;23(2):85-90. doi: 10.1097/YCO.0b013e3283366657. PMID 20061953